CLINICAL TRIAL: NCT03755089
Title: Oral Phenazopyridine Versus Intravesical Lidocaine for Office OnabotulinumtoxinA Analgesia: A Randomized Controlled Trial
Brief Title: Oral vs Intravesical Analgesia for Office Bladder Botox Injections
Acronym: OPIL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1258364-2
Record Dates: First submitted 2018-11-26; First posted 2018-11-27 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Overactive Bladder Syndrome; Urge Incontinence; Urinary Incontinence; Detrusor Hyperreflexia; Detrusor Instability
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Incontinence; Urinary Bladder, Overactive | interventions — Phenazopyridine; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Phenazopyridine (Active Comparator): Patients randomized to the oral phenzopyridine arm will receive 200mg phenazopyridine to take by mouth 1-2 hours before their scheduled procedure.
  Interventions: Drug: Phenazopyridine
- Intravesical Lidocaine (Active Comparator): Patients randomized to the intravesical lidocaine arm will have the bladder back-filled with 30mL 2% lidocaine for the 20 minutes immediately preceding their procedure.
  Interventions: Drug: Lidocaine 2% Injectable Solution

INTERVENTIONS:
Drug: Phenazopyridine — 200mg PO Phenazopyridine taken 1-2 hours prior to the Botox® injection procedure
  Arms: Oral Phenazopyridine
Drug: Lidocaine 2% Injectable Solution — 30mL 2% lidocaine instilled into the bladder lumen 20 via a urinary catheter 20 minutes prior to the Botox® injection procedure
  Arms: Intravesical Lidocaine

SUMMARY:
OnabotulinumtoxinA (Botox®) bladder injections are a highly effective treatment for overactive bladder and urgency urinary incontinence. The procedure is typically performed in the office setting with one of two medications to control comfort. However, the effectiveness of these medications has never been compared. The goal of this study is to determine which medication is better at providing comfort during bladder Botox® injections.

DETAILED DESCRIPTION:
The primary aim of this randomized clinical trial is to compare the analgesic effect of oral phenazopyridine to that of intravesical lidocaine during intradetrusor injections of onabotulinumtoxinA performed for idiopathic overactive bladder. The investigators will achieve this by measuring the mean visual-analog pain scores (VAS) in women who are randomized to receive either oral phenazopyridine or intravesical lidocaine.

Secondary aims include assessment of:

1. Overall Patient Satisfaction: To compare overall patient satisfaction with the onabotulinumtoxinA injection procedure in women randomized to pre-procedure oral phenazopyridine versus those randomized to intravesical lidocaine instillation.
2. Ease of Procedure: To compare the physician's perception of ease of onabotulinumtoxinA injection procedure in women randomized to pre-procedure oral phenazopyridine versus those randomized to intravesical lidocaine instillation.
3. Office Efficiency/Total Appointment Duration: To compare total appointment time or total time spent in an office exam/procedure room in women randomized to pre-procedure oral phenazopyridine versus those randomized to intravesical lidocaine instillation.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant, adult females 18 years of age or older
* Diagnosis of idiopathic overactive bladder
* Planning office-based bladder injection of onabotulinumtoxinA
* Willing and able to complete all study related items and interviews
* Grossly neurologically normal on exam

Exclusion Criteria:

* Known neurologic diseases (multiple sclerosis, Parkinson Disease, CVA within 6 months, myasthenia gravis, Charcot-Marie-Tooth disease, peripheral neuropathy, and complete spinal cord injury) believed to affect urinary function
* Planned injection of >100 units of onabotulinumtoxinA
* OnabotulinumtoxinA given for another indication within the previous 3 months (if cumulative dose would total >400 units)
* Any intradetrusor onabotulinumtoxinA injections in the previous 12 months
* Serum creatinine level greater than twice the upper limit of normal within the year prior to enrollment
* Allergy to lidocaine
* Allergy to onabotulinumtoxinA
* Allergy to phenazopyridine
* Untreated urinary tract infection (UTI)
* Currently pregnant or lactating.
* Known urinary retention (post-void residual >200mL) and inability to perform intermittent self-catheterization
* Uninvestigated hematuria (gross or microscopic)
* Current or prior bladder malignancy
* Previous bladder augmentation or surgically altered detrusor muscle
* Prior pelvic radiation
* Primary language other than English or Spanish

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Analgesic Effect Measured with 100mm Visual Analog Scale | Immediately post-procedure
  The visual analog scale is a visual representation of pain severity rated from 0 (no pain) to 10 (worst pain imaginable). Therefore higher numbers represent more pain.The scale is represented visually using a 100 millimeter line and patients indicate their level of pain by pointing to a location on the line.

SECONDARY OUTCOMES:
Overall Patient Satisfaction | Immediately post-procedure
  Overall patient satisfaction with the onabotulinumtoxinA injection procedure in women randomized to pre-procedure oral phenazopyridine versus those randomized to intravesical lidocaine instillation. Overall satisfaction will be measured with a single-item question utilizing a Likert scale with options ranging from very satisfied to very unsatisfied.
Ease of Procedure | Immediately post-procedure
  Physician's perception of ease of onabotulinumtoxinA injection procedure in women randomized to pre-procedure oral phenazopyridine versus those randomized to intravesical lidocaine instillation. This will be measured with a single item, five point Likert scale with options ranging from no difficulty to great difficulty.
Office Efficiency/Total Appointment Duration | Immediately post-procedure
  Total appointment time or total time spent in an office exam/procedure room in women randomized to pre-procedure oral phenazopyridine versus those randomized to intravesical lidocaine instillation. This will be measured by subtracting the appointment start time (time the patient was placed in the exam room) from the appointment end time (time of patient check-out).

CONTACTS AND LOCATIONS:
Overall Officials: Lauren E Stewart, MD, Principal Investigator — Women and Infants Hospital of Rhode Island
Locations (1):
- Women & Infants Hospital of Rhode Island, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stewart LE, Siddique M, Jacobs KM, Raker CA, Sung VW. Oral phenazopyridine vs intravesical lidocaine for bladder onabotulinumtoxinA analgesia: a randomized controlled trial. Am J Obstet Gynecol. 2022 Aug;227(2):308.e1-308.e8. doi: 10.1016/j.ajog.2022.05.025. Epub 2022 May 14. PMID 35580634